CLINICAL TRIAL: NCT01698580
Title: Effectiveness of a Multifactorial Falls Prevention Program in Community-dwelling Older People When Compared to Usual Care: A Randomized, Controlled Trial
Brief Title: Multifactorial Falls Prevention Program - Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Cidade de Sao Paulo (Other); University of Sao Paulo General Hospital (Other); The George Institute (Other)
Responsible Party: Principal Investigator, Luiz Eugenio Garcez Leme, MD, PhD Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAPPesq 0145/11
Record Dates: First submitted 2012-08-30; First posted 2012-10-03 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Accidental Falls
Keywords: accidental falls; aged; aged, 80 and over; prevention and control

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (Active Comparator): The control group will receive a baseline assessment to identify risk factors for falls and will be referred to their clinicians with a report of individual modifiable risk factors to be managed without any specific guidance: referral to routine services, treatments or any specific orientation will be at the discretion of their primary clinicians. So, further management of each participant in the control group will be individualized, with no specific protocol. Interventions will be recorded. Participants will receive a leaflet with basic orientations for fall prevention.
  Interventions: Other: Usual care
- Multifactorial Falls Prevention Program (Experimental): 12 week intervention for 10 to 12 participants with sessions once a week, lasting for 2 hours, consisting of: On-site exercises (progressive body balance exercise program),Home-based exercise program, Educational and Behavioural sessions and management of modifiable risk factors.
  Interventions: Other: On-site exercise; Other: home-based exercise; Other: Educational and behavioural; Other: Management of modifiable risk factors

INTERVENTIONS:
Other: On-site exercise — The program will consist of progressive balance, including postural orientation and anticipatory postural adjustments sensory-motor activities, and strengthening exercises to enhance balance and postural control and reduce falls. Exercises in the standing position will be prioritised in order to target balance control.Exercises will be both static and dynamic, and will get progressively more challenging, in order to reach the individual optimal level of balance and strength functional status.
  Other Names: balance exercises; strengthening exercises
  Arms: Multifactorial Falls Prevention Program
Other: home-based exercise — Participants will be provided with a detailed booklet containing safety precautions, instructions and photographs of exercises for use in exercise sessions at home and will be instructed to do the exercises preferably under the supervision of a relative or caregiver, in a suitable place (with good lighting and ventilation) and using proper support (close to a table or chair, or the corner of a wall). In the first four weeks of intervention the patients will stay for 30 minutes after the therapy sessions in order to learn the home exercises. The exercises will be reviewed, if necessary, after each session till the last week of intervention. All necessary equipment to undertake the exercise program will be provided.
  Other Names: balance exercises; strengthening exercises
  Arms: Multifactorial Falls Prevention Program
Other: Educational and behavioural — Sessions will address specific environmental and behavioural risk factors delivered by trained health professionals,lasting for 30 minutes and will use appropriate language for lay people.Each meeting will be consisted of a brief introduction on the core day topic with supporting audio-visual or graphic material, followed by group discussion in order to identify the beliefs and attitudes of participants regarding falls and any major restriction or barrier for the implementation of preventive strategies. Participants will be encourage to report their own experiences and beliefs. The activity will always end with the reinforcement of the core message of the session.
  Arms: Multifactorial Falls Prevention Program
Other: Management of modifiable risk factors — Postural hypotension: review of medications that may contribute to postural hypotension;Visual impairment: Participants identified as having visual problems will be referred to an ophthalmologist. The use of four or more medications or the use of psychotropic medication: A review of the risk-benefit of using specific medications will be undertaken, especially psychotropic and anti-hypertensive drugs; Foot problems and shoes: Guidance on the use of proper footwear, nail care and the treatment of cutaneous mycoses will be given; Undernutrition: Participants with a BMI lower than 22 kg / m2 and or a leg calf under 31cm will be oriented to increase their protein and calorie intake and will be referred to a nutritionist.
  Arms: Multifactorial Falls Prevention Program
Other: Usual care — The control group will receive a baseline assessment to identify risk factors for falls and will be referred to their clinicians with a report of individual modifiable risk factors to be managed without any specific guidance: referral to routine services, treatments or any specific orientation will be at the discretion of their primary clinicians. So, further management of each participant in the control group will be individualized, with no specific protocol. Interventions will be recorded. Participants will receive a leaflet with basic orientations for fall prevention.
  Arms: usual care

SUMMARY:
This study is a clinical trial designed to evaluate the effectiveness of a multifactorial falls prevention program in reducing the rate of falls.

A multifactorial falls prevention program consisting of an individualized medical management of the modifiable risk factors, a progressive on-site body balance exercise plus a home-based exercise program, an educational/behavioral intervention and a fall prevention booklet will reduce the number of falls and fall rates when compared with usual care.

DETAILED DESCRIPTION:
This study is a multicenter parallel-group randomized trial among community-dwelling men and women aged 60 years and over, who have fallen at least once in the previous year. Participants will be recruited in multiple settings in Sao Paulo - Brazil and will be randomly allocated to a control group or an intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults, men and women aged 60 and over who have fallen at least once in the last 12 months

Exclusion Criteria:

* A previous diagnosis of dementia or a cognitive decline;
* A previous stroke with a severe neurological impairment;
* A progressive neurological disease;
* A severe visual deficiency;
* Any acute illness that the physician considers as an exercise contra-indication;
* An acute vertigo or dizziness less than 3 months duration;
* Inability to keep on standing, even with the use of a walking aid or other device;
* Unable to communicate;
* Those who are engaged in a regular exercise program, including physical therapy, with a frequency of equal to or more than twice a week such as: muscle strengthening, balance or gait exercise, Tai Chi and Yoga

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2013-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
rate of falls | 12 months
  Participants will receive instructions to fill in a monthly fall diary. They will receive telephone calls each month to ask for information regarding falls and its consequences, such as the mechanisms, environmental conditions, place (indoors or outdoors), activity during the fall and consequences.
proportion of fallers | 12 months
  Participants will receive instructions to fill in a monthly fall diary. They will receive telephone calls each month to ask for information regarding falls and its consequences, such as the mechanisms, environmental conditions, place (indoors or outdoors), activity during the fall and consequences.

SECONDARY OUTCOMES:
Fall-related self-efficacy | baseline, 6 months, 12 months
  will be assessed by the Falls Efficacy Scale International, translated and adapted in its Brazilian version
Balance: Berg Balance Scale, Alternate step test, sit to stand test | baseline, 6 months and 12 months
  Berg Balance Scale Alternate Step Test Sit to stand test
Fall risk: Quick Falls Risk Assessment | baseline, 6 months, 12 months
  Quick Screen Clinical Falls Risk Assessment
The level of difficulty with daily tasks | baseline, 6 months, 12 months
  Brazilian OARS Multidimensional Functional Assessment Questionnaire (BOMFAQ)
Services use | 6 months, 12 months
  number of visits to emergency units, hospitalisation (frequency and time) that each participant will have to treat a fall and or it consequences.
Strength: Grip Strength with a dynamometer | Strength
  Hand grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Perracini, PT, PhD, Principal Investigator — Universidade Cidade de Sao Paulo; Luiz Eugenio G Leme, MD, PhD, Study Director — University of Sao Paulo; Sergio O Paschoal, MD, PhD, Study Chair
Locations (1):
- University of Sao Paulo - Orthopedics Institute, São Paulo, Brazil

REFERENCES:
- [Derived] de Negreiros Cabral K, Perracini MR, Soares AT, de Cristo Stein F, Sera CT, Tiedemann A, Sherrington C, Filho WJ, Paschoal SM. Effectiveness of a multifactorial falls prevention program in community-dwelling older people when compared to usual care: study protocol for a randomised controlled trial (Prevquedas Brazil). BMC Geriatr. 2013 Mar 15;13:27. doi: 10.1186/1471-2318-13-27. PMID 23497000